CLINICAL TRIAL: NCT00169572
Title: See Detailed Description
Brief Title: Study for The Prevention Of Nausea in Cancer Patients Receiving Highly Emetogenic Cisplatin Based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NKV20001
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2010-05-10 (Estimated); Status verified 2010-05

CONDITIONS: Nausea and Vomiting; Chemotherapy-Induced
Keywords: Nausea; Vomiting; Emesis; Chemotherapy-induced Nausea and Vomiting; CINV
MeSH Terms: conditions — Nausea; Vomiting | interventions — Aprepitant; Ondansetron; casopitant; Dexamethasone

INTERVENTIONS:
Drug: Aprepitant
Drug: Ondansetron
Drug: GW679769
Drug: Dexamethasone
  Other Names: Aprepitant; Ondansetron; GW679769

SUMMARY:
This study was designed to assess the safety and efficacy of an investigational agent administered in addition to a standard anti-emetic regimen for the treatment of chemotherapy induced nausea and vomiting.

DETAILED DESCRIPTION:
Phase II Multicentre, Randomised, Double-Blind, Placebo and Active-Controlled, Dose-Ranging, Parallel Group Study of the Safety and Efficacy of The Oral Neurokinin-1 Receptor Antagonist, GW679769 in Combination with Ondansetron Hydrochloride and Dexamethasone for the Prevention of Chemotherapy-Induced Nausea and Vomiting in Cancer Subjects Receiving Highly Emetogenic Cisplatin-based Chemotherapy.

ELIGIBILITY:
Inclusion criteria:

* Willing to provide a written informed consent prior to receiving any study-specific procedures or assessments.
* Diagnosed with a solid malignant tumour and has not previously received chemotherapy.
* Scheduled to receive chemotherapy conducive to regimens outlined in the study protocol.

Exclusion criteria:

* Not received any investigational product within 30 days of enrolment into the study.
* Must not be pregnant.
* Must not be of childbearing potential or is willing to use specific barrier methods outlined in the protocol.
* Must not be scheduled to receive radiation therapy to the abdomen or to the pelvis within seven (7) days prior to starting study medication.
* Must not be currently under treatment for a condition which may cause nausea or vomiting (i.e., active peptic ulcer disease, gastric obstruction).
* Must not have a history of peptic ulcer disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492
Dates: Start 2005-02

PRIMARY OUTCOMES:
The number of subjects who do not experience vomiting, retching or nausea over a 5 day period following the initiation of chemotherapy.

SECONDARY OUTCOMES:
Routine physical exam findings, vital signs, routine clinical laboratory tests, clinical monitoring and/or observation, and adverse events reporting.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (43):
- Argentina (2):
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Buenos Aires
- Austria (2):
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Vienna
- Belgium (4):
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile
- GSK Investigational Site, Zagreb, Croatia
- Czechia (3):
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Prague
- GSK Investigational Site, Shatin, N.T., Hong Kong
- Hungary (2):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Székesfehérvár
- Italy (7):
  - GSK Investigational Site, Benevento, Campania
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Casalpusterlengo (LO), Lombardy
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Perugia, Umbria
- Mexico (2):
  - GSK Investigational Site, Durango, Durango
  - GSK Investigational Site, Mérida, Yucatán
- Netherlands (4):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Arnhem
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Utrecht
- Pakistan (2):
  - GSK Investigational Site, Karachi
  - GSK Investigational Site, Lahore
- GSK Investigational Site, Callao, Provincia Constitucional del Callao, Peru
- Philippines (2):
  - GSK Investigational Site, Quezon City
  - GSK Investigational Site, Taft Avenue, Manila
- Poland (3):
  - GSK Investigational Site, Bydogoszcz
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Poznan
- GSK Investigational Site, Bucharest, Romania
- GSK Investigational Site, Singapore, Singapore
- Slovakia (2):
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Nitra
- Taiwan (2):
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Tao Yuan County